CLINICAL TRIAL: NCT04508478
Title: The Impact of Exercise Training to Patients With Atrial Fibrillation
Brief Title: Exercise Training to Atrial Fibrillation
Acronym: ExAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202007030RINC
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; weight training; aerobic training; cardio-pulmonary function
MeSH Terms: conditions — Atrial Fibrillation | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic training (Experimental)
  Interventions: Behavioral: Aerobic training
- Resistance training (Active Comparator)
  Interventions: Behavioral: Resistance training
- Control (Placebo Comparator)
  Interventions: Behavioral: Control physical exercise

INTERVENTIONS:
Behavioral: Aerobic training — Aerobic training
  Arms: Aerobic training
Behavioral: Resistance training — Resistance training
  Arms: Resistance training
Behavioral: Control physical exercise — Control physical exercise
  Arms: Control

SUMMARY:
To test the impacts of different exercise training programs to the cardiopulmonary function, muscle metabolism, and body mass composition

DETAILED DESCRIPTION:
Atrial fibrillation (AF) has been a global threat due to its increasing incidence and prevalence, and also its potential complications of embolic stroke and heart failure, and therefore has a great impact on life expectancy and quality of life. AF with preserved ventricular function is associated with exercise intolerance, and the effect of physical training had shown to improve life quality and heart function in the population. However, the optimal physical training modalities and intensities are not well studies.

Here we conduct a prospective, randomized, and interventional trial to investigate the effects of different exercise training programs to the burden of AF. We also exploit advanced imaging modalities, including dual x-ray absorptiometry and muscle magnetic resonance, to explore the change of body mass compositions. With this project, we will be able to explore the effects of different physical exercise modalities to the burden of AF and heart function, and also build up a best exercise training program, specific for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal or persistent atrial fibrillation
2. Daily activity below moderate intensity < 300 minutes or high intensity < 150 minutes per week.

Exclusion Criteria:

1. Active infection.
2. Implant cardiac pacemaker.
3. Uncontrolled hypertension.
4. Cardiopulmonary contraindication to exercise training, such as decompensated heart failure, acute pulmonary edema, unstable angina, uncontrolled arrhythmia causing hemodynamic compromise, symptomatic severe aortic stenosis, suspected dissecting aortic aneurysm, severe pulmonary hypertension, acute myocarditis, endocarditis or pericarditis, uncontrolled asthma and SpO2 < 90% at rest on room air.
5. Inability to follow verbal command or to walk on treadmill or use stationary bike.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AF burden | 5 months
  AF burden on 14 day ECＧ
CPET/6 minute walking test | 5 months
  CPET/6 minute walking test
DEXA/muscle MRI | 5 months
  DEXA/muscle MRI

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Yu, MD.PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No